CLINICAL TRIAL: NCT04659018
Title: Development of a Serum Test for Colorectal Cancer Screening
Brief Title: Development of a Serum Test for Colorectal Cancer Screening (COLODIAG préclinique)
Acronym: COLODIAG pre
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MANFREDI Oncodiag 2019
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient: individual performing a screening colonoscopy
  Interventions: Biological: blood collection

INTERVENTIONS:
Biological: blood collection — A 5ml blood sample will be taken in a dry tube when the venous line necessary for the general anaesthesia for the colonoscopy is placed.

SUMMARY:
Colorectal cancer (CRC) is a major public health problem, with 44,872 new cases per year in France (3rd most common cancer), and 17,684 deaths (2nd cause of death from cancer).

Colorectal cancer screening is used to detect early-stage cancers and precancerous lesions (adenomas). Detecting the disease at an early stage enables curative treatment, which is less aggressive and less costly than treatment at an advanced stage.

Fecal occult blood screening has proven its effectiveness in the general population, with a 14% to 16% reduction in colorectal cancer mortality, and even a drop in incidence with 2nd generation immunological tests (FIT).

In France, organised colorectal cancer screening in the general population has been in place since 2009 and since 2015 has been based on the use of a quantitative immunological test (OC-Sensor®).

This test is offered every 2 years to men and women aged between 50 and 74 with an average risk of developing CRC, i.e. nearly 19.7 million people.

The disadvantages of the current screening test are:

* Insufficient sensitivity, although the FIT is more sensitive than the old guaiac test, its sensitivity is not perfect.
* Insufficient specificity: many colonoscopies are performed for nothing. This unjustifiably exposes many patients to endoscopic complications and incurs an unnecessary cost to society.
* The participation rate in screening is too low. Colorectal cancer screening participation was 32.1% in 2017/2018, below the European minimum efficiency target of 45% and far below the 71% observed in our Dutch neighbours.

Several non-invasive alternatives for colorectal cancer screening are being explored and proposed. Among these techniques, serum protein assay has shown its interest in terms of screening for adenomas and colorectal cancers. The assay of 7 serum proteins (which will be the subject of a patent application in 2020), by ELISA test, is the subject of this study.

These results need to be confirmed in a prospective study, with comparison to the gold standard: total colonoscopy. If these results are confirmed, this would make it possible to develop a new non-invasive method of colorectal cancer screening, which would have several advantages over the current test: better sensitivity than the FIT (estimated at about 38% for the detection of advanced adenomas and 88% for colorectal cancers) which would limit the number of false negatives and decrease the number of colorectal cancers discovered at a late stage, a better specificity which would limit the number of false positives and decrease the number of unnecessary colonoscopies, a better participation in the screening test, and a reasonable cost with a technique that can be routinely performed in many centres.

Prior to this prospective clinical study, a pre-clinical calibration phase of the test (combined dosage of the 7 candidate proteins) is necessary, which is the subject of the present project.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given oral consent
* Individual performing a screening colonoscopy either as part of mass screening for colorectal cancer (medium risk, FIT positive) or as part of a personal or family history of adenoma or colorectal cancer (high risk).

Exclusion Criteria:

* A person who is not affiliated with national health insurance
* Person subject to a measure of legal protection (guardianship, tutorship)
* Person subject to a court order
* Pregnant, parturient or breastfeeding woman
* Adult who is unable to provide consent
* Minor
* Individuals at very high risk of colorectal cancer
* Symptomatic individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individual performing a screening colonoscopy either as part of mass screening for colorectal cancer (medium risk, FIT positive) or as part of a personal or family history of adenoma or colorectal cancer (high risk).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
The ability to predict the presence of adenomas and colorectal cancers. | to inclusion
  Development and calibration of the ELISA test measuring the 7 candidate proteins.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France